CLINICAL TRIAL: NCT03406767
Title: A Comparison Between a Standardized (GLA:D Canada) and an Individualized (JointEffort) Exercise Program on Functional Mobility, Quality of Life, Pain Management, and Inflammatory Biomarkers in Knee Osteoarthritis Patients
Brief Title: A Comparison Between GLA:D Canada and an Individualized JointEffort Exercise Program in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: McCaig Institute for Bone and Joint Health (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00077351
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This study involves evaluation of knee osteoarthritis patients who are participating in one of two existing community-based exercise programs (i.e., the GLA:D® or the JointEffort program). Given the pre-experimental design participants will be enrolled after they have registered for one of the two programs (i.e., participants will not be allocated to group assignment) and there is no control group.
  1. The GLA:D® program consists of 1) pre and post program self-reported and functional outcome measures; 2) 2, 1.5 hour education sessions; and 3) neuromuscular exercise training program administered in 1 hour, small (up to 10 persons) group-based, supervised sessions twice weekly for 6 weeks.
  2. The Joint Effort program consists of: 1) one visit aimed at individualized program design; 2) registered dietician led nutrition seminar; and 3) individualized exercise training program administered in 1 hour, small (up to 10 persons) group-based, supervised sessions twice weekly for 6 weeks.
Who Masked: Outcomes Assessor
Masking Description: As both intervention arms are exercise-based it is impossible to mask the participants or individuals delivering the programs.
  All outcome measurements will be performed by a research assistant who is blinded to participant group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLA:D Canada Program (Experimental): GROUP 1: GLA:DTM CANADA GROUP (STANDARDIZED EXERCISE PROGRAM)
  Interventions: Other: GLA:D Canada Program
- JointEffort Program (Experimental): GROUP 2: JOINTEFFORT GROUP (INDIVIDUALIZED EXERCISE PROGRAM)
  Interventions: Other: JointEffort Program

INTERVENTIONS:
Other: GLA:D Canada Program — The GLA:D® program consists of 1) pre- and post-program outcome measurement (self-reported and functional outcomes); 2) 2, 1-1.5 hour education sessions including information on OA disease characteristics, treatments and self-help strategies; and 3) a neuromuscular exercise (warm-up, circuit training, and cool down) training program administered in 1 hour, small (up to 10 persons) group-based, supervised sessions twice weekly for 6 weeks. The goal of the exercises is to restore neutral, functional alignment of the legs by building compensatory functional stability and improving sensorimotor control.
  Arms: GLA:D Canada Program
Other: JointEffort Program — The JointEffort program consists of: 1) one appointment aimed at individualized program design (1-1.5 hours); 2) a nutritional seminar taught by a registered dietician explaining dietary recommendations for OA patients and inflammatory conditions, including weight loss and/or management (1 hours); and 3) an individualized exercise (strength and neuromuscular training, balance training, and range of motion exercises) training program administered in 1 hour, small (up to 10 persons) group-based, supervised sessions twice weekly for 6 weeks.
  Arms: JointEffort Program

SUMMARY:
Osteoarthritis (OA) is the leading cause of disability worldwide and affects more than 4.4 million people in Canada (13% of Canadians). OA symptoms include joint pain, stiffness, range of motion loss, and inflammation, resulting in a significant decrease in quality of life. Current evidence-based guidelines for OA management recommend weight loss, patient education, exercise therapy, bracing, viscosupplementation, and anti-inflammatory/pain medications prior to joint replacement surgery. Unfortunately, current practice trends are not consistent with these guidelines and focus largely on joint replacement. Recently, research from a group in Denmark has shown a reduction in the progression of knee OA symptoms, joint related painkiller use, individuals on sick leave, and higher physical activity levels 12 months after a combined patient education and standardized group exercise therapy program (GLA:D®). Based on the Danish success, the GLA:D® program has been made available in Canada. To date it is unclear if the GLA:DTM Canada program will result in outcomes similar to those seen in Denmark, or how the GLA:DTM program compares to existing individualized OA care programs (i.e. JointEffort). This research will answer the following three questions;

1. Is the GLA:DTM standardized education and exercise program associated with improvements in functional mobility, quality of life, pain management, and inflammatory biomarkers in knee OA patients in Calgary, Alberta?
2. Is the JointEffort individualized exercise and education program associated with improved functional mobility, quality of life, pain management, and inflammatory biomarkers in knee OA patients in Calgary, Alberta?
3. Do the improvements in functional mobility, quality of life, pain management, and inflammatory biomarkers in knee OA patients differ between those enrolled in the GLA:DTM and the JointEffort education and exercise programs?

DETAILED DESCRIPTION:
BACKGROUND:

Osteoarthritis (OA) is the leading cause of disability worldwide and affects more than 4.4 million people in Canada (13% of Canadians). OA symptoms include joint pain, stiffness, range of motion loss, and inflammation, resulting in a significant decrease in quality of life. Current evidence-based guidelines for OA management recommend weight loss, patient education, exercise therapy, bracing, viscosupplementation, and anti-inflammatory/pain medications prior to joint replacement surgery. Unfortunately, current practice trends are not consistent with these guidelines and focus largely on joint replacement. Recently, research from a group in Denmark has shown a reduction in the progression of knee OA symptoms, joint related painkiller use, individuals on sick leave, and higher physical activity levels 12 months after a combined patient education and standardized group exercise therapy program (GLA:D®). Based on the Danish success, the GLA:D® program has been made available in Canada. To date it is unclear if the GLA:D® Canada program will result in outcomes similar to those seen in Denmark, or how the GLA:D® program compares to existing individualized OA care programs (i.e. JointEffort).

RESEARCH QUESTIONS:

1. Is the GLA:D® standardized education and exercise program associated with improvements in functional mobility, quality of life, pain management, and biomarkers in knee OA patients in Alberta?
2. Is the JointEffort individualized exercise and education program associated with improved functional mobility, quality of life, pain management, and biomarkers in knee OA patients in Alberta?
3. Do the improvements in functional mobility, quality of life, pain management, and biomarkers in knee OA patients differ between those enrolled in the GLA:D® and the JointEffort education and exercise programs?

OBJECTIVES:

The objectives of this pre-experimental intervention study are to 1) assess the association between participation in the GLA:D® standardized program and functional mobility, quality of life, pain management, and inflammatory biomarkers in knee OA patients, 2) assess the association between participation in the JointEffort individualized program and functional mobility, quality of life, pain management, and inflammatory biomarkers in knee OA patients, and 3) assess if there are any differences in outcomes between the standardized (GLA:D®) and individualized (JointEffort) exercise programs.

METHODOLOGY:

Study Participants: A convenience sample of 60 participants ≥50 years of age with a primary care physician or orthopedic surgeon knee OA diagnosis will be included in the study. Specifically, 30 individuals will participate in 1) the GLA:D® program and 30 sex- and age-matched individuals will participate in 2) the JointEffort program. 60 participants is a conservative estimate based on the ability to detect a moderate effect between study groups (1-β=0.8, α=0.05).

Exercise Programs: The GLA:D® program consists of 1) pre- and post-program outcome measurement (self-reported and functional outcomes); 2) 2, 1-1.5 hour education sessions including information on OA disease characteristics, treatments and self-help strategies; and 3) a neuromuscular exercise (warm-up, circuit training, and cool down) training program administered in 1 hour, small (up to 10 persons) group-based, supervised sessions twice weekly for 6 weeks. The goal of the exercises is to restore neutral, functional alignment of the legs by building compensatory functional stability and improving sensorimotor control. The JointEffort program consists of: 1) one appointment aimed at individualized program design; 2) a nutritional seminar taught by a registered dietician explaining dietary recommendations for OA patients and inflammatory conditions, including weight loss and/or management; and 3) an individualized exercise (strength and neuromuscular training, balance training, and range of motion exercises) training program administered in 1 hour, small (up to 10 persons) group-based, supervised sessions twice weekly for 6 weeks.

Study Outcomes:

1. Demographic (age, sex, height, weight, and body mass index), comorbidity, attendance, exercise log, and medication use details will be recorded at each visit. Adherence will be measured by exercise program attendance (number of sessions).
2. The following self-report questionnaires will be completed at baseline, 2, and 12 months: the Knee Injury and Osteoarthritis Outcome Score (KOOS), the Intermittent and Constant Osteoarthritis Pain (ICOAP) Score, and the EuroQOL-5 Dimensions-5 Levels (EQ-5D-5L) Score.
3. The patient knowledge questionnaire on OA (PKQ-OA) and the arthritis self-efficacy questionnaire will be completed at baseline, 2, and 12 months.
4. All participants will complete the 40m Face-Paced Walk Test and the 30s Chair Stand Test at baseline, 2, and 12 months.
5. A blood serum sample, collected at baseline, 2, and 12 months will be analyzed to assess for biomarkers (cytokines, chemokines, adipokines, mytokines) using a Discovery Assay (42 Custom-Plex human assay) with Luminex-xMAP technology (Eve Technologies).

STATISTICAL ANALYSIS:

Descriptive statistics (mean (95% CI), proportion (95% CI) or median (range) will be used report the baseline, 2, and 12 month change in self-report, functional and biomarker outcomes, as appropriate. To account for the matched design, mean within-pair difference (95% CI) will be used to compare treatment groups across outcomes. Finally, conditional logistic regression will be used to assess the relationship between attendance (number of sessions) and 12-month change in each outcome.

SIGNIFICANCE:

This project will contribute to the understanding of exercise programming prescription for knee OA patients. If GLA:D® and/or JointEffort support improvements in functional mobility, quality of life, pain management, and biomarkers, it could play a role in the implementation strategy for OA patients within the province. Exercise programming has the potential to be implemented in several sites across Alberta, and thus potentially modifying disease progression and possibly delaying total joint replacement.

ELIGIBILITY:
Inclusion Criteria:

1. have been diagnosed with OA by a primary care physician or orthopedic surgeon;
2. ≥50 years of age;
3. are able read, understand, and provide informed consent in English; and
4. can attend exercise programming classes at the University of Calgary.

Exclusion Criteria:

1. have physical or neurological impairments or pre-existing medical conditions where physical activity is contraindicated;
2. have inflammatory arthritis, a fracture, tumor, or acute trauma; and
3. participated in the JointEffort or GLA:D program previously.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) self-report questionnaire | Baseline, 2 and 12 months
  The KOOS self-report questionnaire [17] will be used to evaluate changes in symptoms and function related to knee OA at baseline, 2 and 12 months. Changes from baseline will be reported. The KOOS consists of 42 items in five subscales (pain, other symptoms, function in daily living, function in sport and recreation, and knee-related quality of life) scored on a 5-point Likert scale. Subscale scores will be summed and the total score transformed to a 0-100 scale with higher scores indicating better function.

SECONDARY OUTCOMES:
40m Fast Paced Walk Test | Baseline, 2 and 12 months
  After a practice trial all participants will complete the 40m Face-Paced Walk Test at baseline, 2, and 12 months to provide a measure of physical function (endurance). Changes from baseline will be reported. Participants are asked to walk as quickly but as safely as possible, without running, along a 10 m (33 ft) walkway and then turn around a cone, return then repeat again for a total distance of 40 m (132 ft) (3 turns). If a regular walking aid is needed it will be allowed and its use recorded. The time of trial will be recorded (nearest 100th of a second) and expressed as speed m/s by dividing distance (40m) by time (s).
30 Second Chair Stand Physical Function (Strength) | Baseline, 2 and 12 months
  After a practice trial all participants will complete the 30s Chair Stand Test [13] at baseline, 2, and 12 months to provide a measure of physical function (strength). Changes from baseline will be reported. From a sitting position, on a chair of standardized height each participant will stand up until their hips and knees are fully extended, then sit completely back down, so that their bottom fully touches the seat. This will be repeated for 30 seconds. The number of full sit-to-stand movements in 30 seconds will be recorded. Participant are allowed to stop and rest if they become tired although the time keeps going. If a participant cannot stand even once then the score for the test is zero.
Serum Biomarkers | Baseline, 2 and 12 months
  A blood serum sample, collected at baseline, 2, and 12 months will be analyzed to assess for biomarkers (reported in picograms/ml) using a Discovery Assay (Custom-Plex human assay) with Luminex-xMAP technology (Eve Technologies). Changes from baseline will be reported.
  The biomarkers include the following:
  1. Human Cytokine Array / Chemokine Array.
  2. Human Adipokine Array.
  3. Human Myokine Array.
Arthritis-Related Self-Efficacy Scale | Baseline, 2 and 12 months
  The self-report Arthritis-Related Self-Efficacy Scale will be used to measure patients' arthritis-specific self-efficacy, or patients' beliefs that they could perform specific tasks or behaviors to cope with the consequences of arthritis at baseline, 2 and 12 months. Changes from baseline will be reported. The scale consists of 20 items in 3 subscales(i.e., self-efficacy for managing pain, self-efficacy for physical function, and self-efficacy for controlling other symptoms) scored on a 10-point Likert Scale from very uncertain (1) to very certain (10).
EuroQOL-5 Dimensions self-report questionnaire | Baseline, 2 and 12 months
  The EuroQOL-5 Dimensions (EQ-5D-5L) self-report questionnaire [19] will be used to assess pain, other symptoms, function in daily living, function in sport and recreation, and knee related quality of life at baseline, 2 and 12 months. Changes from baseline will be reported. The EQ-5D-5L consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with 5 response levels from no problems with item (1) to unable to perform item (5), in addition to a percentage score of overall perceived health.
Intermittent and Constant Osteoarthritis Pain self-report questionnaire | Baseline, 2 and 12 months
  The Intermittent and Constant Osteoarthritis Pain (ICOAP) self-report questionnaire [20] will be used to assess pain, taking into account both constant and intermittent pain experiences at baseline, 2 and 12 months. Changes from baseline will be reported.The 11-item tool is divided into 2 subscales: 1) constant pain (intensity, affected sleep, quality of life disruption, frustration and worrying about knee pain) and 2) pain that comes and goes (intensity, frequency, affected sleep, quality of life disruption, and frustration and worrying about knee pain), , each with 5 response levels from no pain (0) to extremely (4).

OTHER OUTCOMES:
Participant Sex | Baseline
  Participants will record their current sex on a custom study questionnaire at baseline. Options will be either male or female.
Participant Age | Baseline, 2 and 12 months
  Participants will record their current age on a custom study questionnaire at baseline, 2 and 12 months.
Participant Height | Baseline, 2 and 12 months
  Participants height will be measured and recorded to the nearest 0.1cm using a standardized stadiometer at baseline, 2 and 12 months.
Participant Weight | Baseline, 2 and 12 months
  Participants weight will be measured and recorded to the nearest 0.1kg using a standardized portable medical scale at baseline, 2 and 12 months.
Participant Body Mass Index (BMI) | Baseline, 2 and 12 months
  BMI will be calculated (kg/m2) and converted into age and sex-specific percentiles using US growth charts, from height (nearest 0.1 cm using a stadiometer) and weight (nearest 0.1 kg using a portable medical scale) measurements.
Participant Medical Comorbidities | Baseline, 2 and 12 months
  Participants will record any current medical comorbidities on a custom study questionnaire at baseline, 2 and 12 months.
Intervention Adherence | Two visits per week over the six weeks of the intervention
  Exercise logs will be recorded at each visit
Medication Use | Baseline, daily over the six week intervention, 2 and 12 months
  Medication use will be logged daily and reviewed with research personnel at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Jackie L Whittaker, PT, PhD, Principal Investigator — Faculty of Rehabilitation Medicine, University of Alberta
Locations (4):
- Canada (4):
  - McCaig Institute for Bone and Joint Health, University of Calgary, Calgary, Alberta
  - Active Living, University of Calgary, Calgary, Alberta
  - Sports Medicine Centre, University of Calgary, Calgary, Alberta
  - Department of Physical Therapy, Faculty of Rehabilitation Medicine, University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of data with other researchers.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03406767/Prot_SAP_002.pdf
  • Informed Consent Form (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03406767/ICF_003.pdf